CLINICAL TRIAL: NCT07386964
Title: Radicle Clarity CNM™: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes Among E-Gamers
Brief Title: Radicle Clarity CNM™: A Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes Among E-Gamers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_P_2606_CNM
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Function

STUDY DESIGN:
Intervention Model Description: Eligible participants must complete all enrollment steps to be stratified. Participants will be stratified based on their sex assignment at birth and health outcome score during enrollment, and e-gamer status, then randomized to one of the study groups sequentially based on all stratification measures collectively to ensure equal distribution to each study product group. Participants will be provided the study product and an insert with additional information on product usage and study procedures.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Clarity Control (Placebo Comparator): Clarity Product Placebo Control
  Interventions: Dietary Supplement: Clarity Product Placebo Control
- Active Clarity Product (Experimental): Clarity Active Product
  Interventions: Dietary Supplement: Clarity Active Product

INTERVENTIONS:
Dietary Supplement: Clarity Product Placebo Control — Participants will use their Clarity Product Placebo Control as directed for a period of 8 weeks
  Arms: Placebo Clarity Control
Dietary Supplement: Clarity Active Product — Participants will use their Clarity Active Product as directed for a period of 8 weeks
  Arms: Active Clarity Product

SUMMARY:
Radicle Clarity CNM™: A randomized, double-blind, placebo-controlled direct-to-consumer study assessing the impact of health and wellness products on cognitive function and related health outcomes among E-Gamers.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants (1) are aged 21-45, (2) either young professionals or e-gamers, (3) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (4) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 9 weeks. Participant reports of health indicators will be collected at enrollment and throughout the active period of study product usage. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion

Participants must meet all the following criteria:

* Adults, aged 21 - 45 years at the time of electronic consent, inclusive of all ethnicities, races, and gender identities

  * Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Identifies as a young professional (working 30+ hrs/week)
* May identify as an E-gamer (playing video games 5+hrs/week for the past year)
* Resides in the United States
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion

Individuals who report any of the following during screening may be excluded from participation:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English at a 7th grade level
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  * NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | 9 weeks
  Change in cognitive function: Difference in rates of change over time in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where lower scores correspond to worse cognitive function)

SECONDARY OUTCOMES:
Change in cognitive abilities | 9 weeks
  Change in cognitive abilities: Difference between rates of change over time in Cognitive Abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)
Change in fatigue | 9 weeks
  Change in fatigue: Difference in rates of change over time in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)

OTHER OUTCOMES:
Minimal clinically important difference (MCID) in cognitive function | 9 weeks
  Minimal clinically important difference (MCID) in cognitive function: Likelihood of experiencing minimal clinically important difference in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where lower scores correspond to worse cognitive function)
Minimal clinically important difference (MCID) in cognitive abilities | 9 weeks
  Minimal clinically important difference (MCID) in cognitive abilities: Likelihood of experiencing minimal clinically important difference in cognitive abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)
Minimal clinically important difference (MCID) in fatigue | 9 weeks
  Minimal clinically important difference (MCID) in fatigue: Likelihood of experiencing minimal clinically important difference in fatigue score as assessed by PROMIS Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com